CLINICAL TRIAL: NCT04048889
Title: Addition of Popliteal Plexus Block to Continuous Femoral Nerve Block for Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Kevin Stebler, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-00655
Record Dates: First submitted 2019-07-27; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized controlled triple-blinded trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal plexus block and continuous femoral nerve block (Experimental)
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- continuous femoral nerve block (Active Comparator)
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Continuous femoral nerve block with injection of 15 mls of Ropivacain 0.5% adjacent to the lateral aspect of the femoral nerve below the fascia iliaca and placement of the catheter within the vicinity of the femoral nerve, juste deep to the fascia iliaca
  Other Names: Continous femoral nerve block
  Arms: continuous femoral nerve block
Drug: Ropivacaine 0.5% Injectable Solution — Continuous femoral nerve block with injection of 15 mls of Ropivacain 0.5% adjacent to the lateral aspect of the femoral nerve below the fascia iliaca and placement of the catheter within the vicinity of the femoral nerve, juste deep to the fascia iliaca.
  Other Names: Continous femoral nerve block
  Arms: Popliteal plexus block and continuous femoral nerve block
Drug: Ropivacaine 0.5% Injectable Solution — Popliteal plexus block with injection of 15 mls of Ropivacain 0.5% inside the distal end of the adductor canal close to the adductor hiatus, adjacent to the femoral artery, between the medial vastus muscle and the adductor Magnus muscle, done under general anesthesia.
  Other Names: Popliteal plexus block
  Arms: Popliteal plexus block and continuous femoral nerve block

SUMMARY:
The popliteal plexus block has been described as an alternative analgesic postoperative pain treatment for total knee arthroplasty. It consists of injecting local anaeshetics inside the distal end of the adductor canal close to the adductor hiatus, adjacent to the femoral artery, between the medial vastus muscle and the adductor magnus muscle, in order to anesthetize the popliteal plexus. However, the analgesic efficacy has never been demonstrated in a randomized controlled trial. Therefore the objective of this study is to investigate the analgesic benefit of this block combined with a continuous femoral nerve block, on patients scheduled for total knee athroplasty.

DETAILED DESCRIPTION:
Patients scheduled to undergo total knee arthroplasty under general anesthesia will be randomly allocated to two groups: continuous femoral nerve block alone or continuous femoral nerve block with addition of a popliteal plexus block.

The continuous femoral nerve block will be performed by the anesthesiologist with 15 mLs of ropivacaine 0.5%, under ultrasound guidance before the beginning of the general anesthesia. The popliteal plexus block will be done by the anesthesiology, under ultrasound guidance, before the beginning of the surgery, under general anesthesia.

Postoperative analgesia will include acetaminophen (4 x 1000 mg), ibuprofen (3 x 400 mg) and a continuous infusion of Ropivacaine 0.2%.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee athroplasty under general anesthesia
* ASA 1-3

Exclusion Criteria:

* Kidney disease with GFR < 50 ml/mn
* Daily opioid consumption > 1 month
* Allergy to local anesthetics
* Neurological problems of the lower extremity
* other contraindications to peripheral nerve blocks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Total iv morphine consumption (mg) | 12 postoperative hours

SECONDARY OUTCOMES:
Total iv morphine consumption (mg) | 24 and 48 postoperative hours
Average and maximum pain scores (Numeric rating scale 0-10) | 12, 24 and 48 postoperative hours
Sciatic extension of popliteal plexus block | 2 and 24 postoperative hours
  Presence of sensitive or/and motor sciatic extension of popliteal plexus block
Plantarflexion and dorsiflexion ankle strength (Newtons) | 2 and 24 postoperative hours
Knee pain localization (anterior, internal, posterior, lateral, medial) | 2, 12, 24 and 48 postoperative hours
Popliteal plexus block procedure time (minutes) | When performing the popliteal plexus block
  Onset of action = beginning of the disinfection; End of action = end of injection of 15 mls of Ropivacain 0.5%
Popliteal plexus block duration of action (hours) | up to 48 postoperative hours
  Onset of action = Time from end of infection of 15 mls of Ropivacain 0.5%; End of action = onset of lateral and/or posterior knee pain (With Numeric rating scale ≥ 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Anesthesia, Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stebler K, Elia N, Zaccaria I, Fournier RM. Popliteal plexus block in total knee arthroplasty: a single-center randomized controlled double-blinded trial. Reg Anesth Pain Med. 2024 Dec 20:rapm-2024-105782. doi: 10.1136/rapm-2024-105782. Online ahead of print. PMID 39709189